CLINICAL TRIAL: NCT07080736
Title: Evaluation of E-learning on Suicide Prevention for Professionals in a Detention Context
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2025-0183
Record Dates: First submitted 2025-06-20; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): Once participants have given their consent online, they receive the first questionnaire. Once this questionnaire is completed, a link to the e-learning is provided. Participants then receive an invitation to complete the post-test. The measurements thus take place just before getting the formation (pretest) and after the formation (post-test). After three days, participants receive a reminder e-mail to complete the post-measurement which they can ignore if they have already completed it.
  Interventions: Behavioral: E-learning

INTERVENTIONS:
Behavioral: E-learning — The training consists of an e-learning module created on the RISE - Articulate platform, and is based on previously developed e-learning modules (SP-reflex) and physical training aimed at other target groups, but was adapted to the specific context of detention.
  This specific training will consist of sensitising information, theoretical knowledge, as well as some concrete tools and tips for suicide prevention within detention. Relevant examples and cases will be discussed. The following topics, among others, will be discussed:
  * How common is suicide?
  * What myths exist about suicide?
  * Why do people contemplate suicide?
  * What is the process from suicidal thoughts to suicide?
  * How do I recognise signs of suicidal thoughts?
  * What can I do if I notice signs?
  * What if someone attempts suicide or a suicide occurs?
  * How do I take care of myself?

SUMMARY:
This study aims to investigate to what extent a gatekeeper training (e-learning) for people working in prison is applicable in their daily practice.

Moreover the study wants to investigate the impact of the e-learning on the knowledge, the attitudes and perceptions of the people working in prison on suiicide (prevention) as well as their feeling of self-efficacy in dealing with people in prison suffering from suicidal ideation of behavior.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years old Have access to internet Speak Dutch Working within a penitentiary institution, in particular in the establishments in Ypres, Merksplas, Bruges and Mechelen.

Exclusion Criteria:

Staff of prisons not working in participating institutions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Applicability | Post test (i.e., immediatly after e-learning of 60-90 minutes); assessed up to 3 days after pre-test
  The primary objective of this study is to evaluate the e-learning module based on participants' perceptions. Specifically, it examines how prison staff assess the content, usability and practicality of the e-learning module. This evaluation provides insight into the extent to which the module meets the needs of the target group and the extent to which it is perceived as relevant and applicable in daily practice.
  Applicability is measured using a self-developed 4-item questionnaire.

SECONDARY OUTCOMES:
Attitudes | Change from Baseline (before e-learning) to post-test (immediatly after e-learning of 60-90 minutes); assessed up to 3 days after pre-test
  Attitudes are measured using the 15-item version of the Attitudes Toward Suicide Scale (ATTS; Renberg & Jacobsson, 2003). Participants respond to 15 statements using a 5-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). The scale assesses various dimensions of participants' attitudes toward suicide.
Self-efficacy | Change from Baseline (before e-learning) to post-test (immediatly after e-learning of 60-90 minutes); assessed up to 3 days after pre-test
  Gatekeeper Self Efficacy Scale (GKSES, Takahashi et al, 2020)is a 9-item self-report questionnaire designed to assess an individual's confidence in their ability to act as a suicide prevention gatekeeper. Each item is rated on a 7-point Likert scale ranging from 1 (Not at all confident) to 7 (Extremely confident), resulting in a total score ranging from 9 to 63.
  Higher scores indicate greater self-efficacy, which reflects a more favorable outcome in terms of perceived gatekeeper competence.

OTHER OUTCOMES:
Sociodemographic information | Baseline (i.e., before the e-learning)
  Participants will be asked to provide basic demographic and professional background information, including age, sex, gender identity, years of work experience, and type of institution of employment (6 items in total).
Experience in suicide (prevention) | Baseline (i.e., before the e-learning)
  Participants report prior experience related to suicide and suicide prevention, including previous training, encounters with suicidal behavior in the prison setting, self-rated level of experience, and knowledge of appropriate referral pathways. This is assessed using 6 self-developed items.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No